CLINICAL TRIAL: NCT01600755
Title: A Prospective Nonrandomized Study of Autologous Muscle Derived Cell (AMDC) Transplantation for Treatment of Fecal Incontinence
Brief Title: Autologous Cell Therapy for Treatment of Fecal Incontinence
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Cook MyoSite (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 09-025
Record Dates: First submitted 2012-05-11; First posted 2012-05-17 (Estimated); Results first posted 2024-02-16 (Actual); Last update posted 2024-02-16 (Actual); Status verified 2023-06

CONDITIONS: Fecal Incontinence
Keywords: Cell Therapy; Autologous Cell Transplantation; Muscle-derived Cell; Anal Incontinence; Rectal Diseases; Intestinal Diseases; Gastrointestinal Diseases; Urinary Incontinence
MeSH Terms: conditions — Fecal Incontinence; Encopresis; Rectal Diseases; Intestinal Diseases; Gastrointestinal Diseases; Urinary Incontinence

ARMS (1):
- Iltamiocel (Experimental): AMDC is the study product (autologous muscle-derived cells). The generic name is iltamiocel. Single intrasphincteric injection of 250 x 10^6 cells.
  Interventions: Biological: Iltamiocel

INTERVENTIONS:
Biological: Iltamiocel — Single intrasphincteric injection of iltamiocel at a dose of 250 x 10^6 cells
  Other Names: Autologous Muscle-Derived Cells (AMDC)

SUMMARY:
The aim of this clinical study is to investigate the safety and feasibility of Autologous Muscle Derived Cells (AMDC, generic name iltamiocel, preparation of a patient's own cells) injection into the anal sphincter for treatment of patients with fecal incontinence.

DETAILED DESCRIPTION:
This study is designed to test the safety and feasibility of iltamiocel (Autologous Muscle Derived Cells, AMDC) as a treatment for fecal incontinence in men and women. Iltamiocel therapy seeks to allow remodeling of the external anal sphincter in patients with fecal incontinence from either defined structural defects or a generalized weakening of the external anal sphincter.

ELIGIBILITY:
Inclusion Criteria:

* Primary symptoms of fecal incontinence, as confirmed by patient medical history and physical examination
* Wexner (Cleveland Clinic Incontinence Severity (CCIS)) score ≥ 9
* Etiology of fecal incontinence is related, at least in part, to external anal sphincter dysfunction
* Failed conservative treatment

Exclusion Criteria:

* Gracilis sling repair or insertion of an artificial sphincter
* Inflammatory Bowel Disease
* Significant rectocele or rectal prolapse
* History of radiation treatment to the anal sphincter or adjacent structures
* Less than 18 years of age
* Pregnant, breastfeeding, or plans to become pregnant during the course of the study
* Neuromuscular disorder
* History of neoplasia within 5 years prior to enrollment, except for basal cell carcinoma, or is receiving or planning to receive anti-cancer medications
* Known bleeding diathesis or uncorrected coagulopathy
* Medical condition that would preclude treatment due to contraindications and/or warnings of concomitant medications or listed in the experimental product labeling
* Compromised immune system due to disease state, chronic corticosteroid use, or other immunosuppressive therapy
* Participating in another investigational drug or device study
* Unable or unwilling to provide informed consent
* Unable or unwilling to commit to the follow-up procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2013-03-28 (Actual); Primary Completion 2021-10-27 (Actual); Study Completion 2021-10-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Manoj J Raval, MD, Principal Investigator — St. Paul's Hospital
Locations (2):
- St. Paul's Hospital, Vancouver, British Columbia, Canada
- Royal London Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Knowles CH, Canestrari E, Jankowski RJ, Cardello K, Raval MJ. Safety and Efficacy of Iltamiocel Cellular Therapy for the Treatment of Fecal Incontinence. Results of a Phase 1/2 Study. Ann Surg. 2023 Dec 1;278(6):937-944. doi: 10.1097/SLA.0000000000005894. Epub 2023 May 5. PMID 37144409

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Iltamiocel
Started | 53
Iltamiocel Injection | 48
3-Month Follow-Up | 48
6-Month Follow-Up | 48
12-Month Follow-Up | 47
Completed | 47
Not Completed | 6
Not completed — Withdrawal by Subject | 6

BASELINE CHARACTERISTICS:
Arm/Group | Iltamiocel
Number analyzed (Participants) | 48
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 24
  >=65 years | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.7 (13.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 47
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 44
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Canada | 33
  United Kingdom | 15
28-Day Incontinence Diary (Number of Episodes) [Median (Full Range); unit: Incontinence Episodes/28 Days] | 16 [0 to 92]
28-Day Incontinence Diary (Days with Episodes) [Median (Full Range); unit: Days with incontinence episodes] | 12 [0 to 28]
Cleveland Clinic Incontinence Score (CCIS) [Mean (Standard Deviation); unit: scores on scales] — CCIS is a validated 5-questions tool assessing the frequency and the type of incontinence episodes (solid, liquid, gas), pad use, and lifestyle alteration. Scored from 0 to 20, with lower scores indicating less severe symptoms.
  scores on scales | 13.6 (2.9)
Fecal Incontinence Quality of Life (FIQL) Questionnaire [Mean (Standard Deviation); unit: scores on scales] — FIQL is a validated, 29-item tool assessing quality of life (QOL) of subjects with FI with four scales: Lifestyle (10 items, scored 0 to 4, with higher scores indicating a better QOL), Coping/Behavior (9 items, scored 0 to 4, with higher scores indicating a better QOL), Depression/Self-Perception (7 items, scored 0 to 4, with higher scores indicating a better QOL), and Embarrassment (3 items, scored 0 to 4, with higher scores indicating a better QOL).
  scores on scales
    FIQL - Lifestyle scale | 2.5 (0.9)
    FIQL - Coping/behavior scale | 1.7 (0.6)
    FIQL - Depression/perception scale | 2.5 (0.9)
    FIQL - Embarrassment scale | 1.9 (0.8)

OUTCOME MEASURES:

1. Primary Outcome: Number of Treatment-Related Adverse Events
Description: Assessment of frequency and severity of adverse events related to study product and study procedures through 12 months following treatment of FI in adult male and female subjects.
Time Frame: 12 months
Measure: Number; unit: events
Arm/Group | Iltamiocel
Number analyzed (Participants) | 53
events
  Study Product-related serious adverse events | 0
  Study Product-related adverse events | 1
  Injection procedure-related adverse events | 5
  Biopsy procedure-related adverse events | 28

2. Secondary Outcome: Number of Fecal Incontinence (FI) Episodes (Median 28-day Fecal Incontinence Diary)
Description: Median number of fecal incontinence (FI) episodes as assessed by 28-day FI diary.
Time Frame: 3, 6, and 12 months post-treatment
Measure: Median (Full Range); unit: Incontinence Episodes/28 Days
Arm/Group | Iltamiocel
Number analyzed (Participants) | 48
Incontinence Episodes/28 Days
  Fecal incontinence diary at 3 months | 8 [0 to 100]
  Fecal incontinence diary at 6 months | 10 [0 to 206]
  Fecal incontinence diary at 12 months | 7 [0 to 161]

3. Secondary Outcome: Number of Days With FI Episodes (Median 28-day Fecal Incontinence Diary)
Description: Median number of days with fecal incontinence (FI) episodes, as assessed by 28-day FI diary.
Time Frame: 3, 6, and 12 months post-treatment
Measure: Median (Full Range); unit: days with incontinence episodes
Arm/Group | Iltamiocel
Number analyzed (Participants) | 48
days with incontinence episodes
  FI diary at 3 months | 7 [0 to 28]
  FI diary at 6 months | 7 [0 to 28]
  FI diary at 12 months | 5 [0 to 28]

4. Secondary Outcome: Number of Participants With Categorical ≥50% Reduction in 28-day Fecal Incontinence Episodes
Description: Number of participants with categorical ≥50% reduction in fecal incontinence (FI) episodes as assessed by 28-day FI diary.
Time Frame: 3, 6, and 12 months post-treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Iltamiocel
Number analyzed (Participants) | 48
Participants
  Fecal incontinence diary at 3 months | 17
  Fecal incontinence diary at 6 months | 19
  Fecal incontinence diary at 12 months | 22

5. Secondary Outcome: Number of Participants With Categorical ≥75% Reduction in 28-day Fecal Incontinence Episodes
Description: Number of participants with categorical ≥75% reduction in fecal incontinence (FI) episodes as assessed by 28-day FI diary.
Time Frame: 3, 6, and 12 months post-treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Iltamiocel
Number analyzed (Participants) | 48
Participants
  Fecal incontinence diary at 3 months | 7
  Fecal incontinence diary at 6 months | 12
  Fecal incontinence diary at 12 months | 16

6. Secondary Outcome: Number of Participants With 100% Reduction in 28-day Fecal Incontinence Episodes
Description: Number of participants with 100% reduction in fecal incontinence (FI) episodes as assessed by 28-day FI diary.
Time Frame: 3, 6, and 12 months post-treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Iltamiocel
Number analyzed (Participants) | 48
Participants
  Fecal incontinence diary at 3 months | 1
  Fecal incontinence diary at 6 months | 4
  Fecal incontinence diary at 12 months | 10

7. Secondary Outcome: Change From Baseline in Patient-reported Quality of Life (Fecal Incontinence Quality of Life (FIQL) Questionnaire)
Description: Mean change from baseline in patient-reported quality of life, as assessed by the Fecal Incontinence Quality of Life (FIQL) questionnaire. The FIQL is a validated, 29-item tool assessing the quality of life (QOL) of subjects with FI with four scales: Lifestyle (10 items, scored 0 to 4, with higher scores indicating a better QOL), Coping/Behavior (9 items, scored 0 to 4, with higher scores indicating a better QOL), Depression/Self-Perception (7 items, scored 0 to 4, with higher scores indicating a better QOL), and Embarrassment (3 items, scored 0 to 4, with higher scores indicating a better QOL).
Time Frame: 3, 6, and 12 months post-treatment
Measure: Mean (Standard Deviation); unit: scores on scales
Arm/Group | Iltamiocel
Number analyzed (Participants) | 48
scores on scales
  Change in FIQL Lifestyle scale at 3 months | 0.4 (0.7)
  Change in FIQL Lifestyle scale at 6 months | 0.4 (0.7)
  Change in FIQL Lifestyle scale at 12 months | 0.6 (0.7)
  Change in FIQL Coping/Behavior scale at 3 months | 0.4 (0.7)
  Change in FIQL Coping/Behavior scale at 6 months | 0.5 (0.7)
  Change in FIQL Coping/Behavior scale at 12 months | 0.5 (0.7)
  Change in FIQL Depression/Self Perception scale at 3 months | 0.3 (0.7)
  Change in FIQL Depression/Self Perception scale at 6 months | 0.3 (0.6)
  Change in FIQL Depression/Self Perception scale at 12 months | 0.4 (0.6)
  Change in FIQL Embarrassment scale at 3 months | 0.5 (0.8)
  Change in FIQL Embarrassment scale at 6 months | 0.5 (0.8)
  Change in FIQL Embarrassment scale at 12 months | 0.6 (0.9)

8. Secondary Outcome: Change From Baseline in Patient-reported Fecal Incontinence Symptom Severity (Cleveland Clinic Incontinence Score (CCIS))
Description: Mean change from baseline in patient-reported fecal incontinence symptom severity, as assessed by the Cleveland Clinic Incontinence Score (CCIS) questionnaire. CCIS is a validated 5-questions tool assessing the frequency and the type of incontinence episodes (solid, liquid, gas), pad use, and lifestyle alteration. Scored from 0 to 20, with lower scores indicating less severe symptoms.
Time Frame: 3, 6, and 12 months post-treatment
Measure: Mean (Standard Deviation); unit: scores on scales
Arm/Group | Iltamiocel
Number analyzed (Participants) | 48
scores on scales
  Change in CCIS score at 3 months | -2.2 (3.0)
  Change in CCIS score at 6 months | -2.0 (2.8)
  Change in CCIS score at 12 months | -2.9 (2.8)

ADVERSE EVENTS:
Time Frame: 12 months
Description: Collection at baseline, 1 month, 3 months, 6 months and 12 months post-treatment
Arm/Group | Iltamiocel
All-Cause Mortality (participants affected / at risk) | 0/53
Serious Adverse Events (participants affected / at risk) | 4/53
Other Adverse Events (participants affected / at risk) | 31/53
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Iltamiocel (N=53)
Pneumonia (Infections and infestations) | 2 (3)
Urinary tract infection (Infections and infestations) | 1 (2)
Urosepsis (Infections and infestations) | 1 (2)
Nephrotic syndrome (Renal and urinary disorders) | 1 (1)
Sinus operation (Surgical and medical procedures) | 1 (1)
Small intestine obstruction (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Iltamiocel (N=53)
Diarrhea (Gastrointestinal disorders) | 8 (9)
Hemorrhoids (Gastrointestinal disorders) | 3 (3)
Proctalgia (Gastrointestinal disorders) | 3 (4)
Cystitis (Infections and infestations) | 3 (4)
Lower respiratory tract infection (Infections and infestations) | 6 (6)
Nasopharyngitis (Infections and infestations) | 4 (4)
Urinary tract infection (Infections and infestations) | 5 (7)
Post procedural contusion (Injury, poisoning and procedural complications) | 5 (5)
Procedural pain (Injury, poisoning and procedural complications) | 14 (14)
Hypoesthesia (Nervous system disorders) | 5 (5)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 30 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication unless confidential information is disclosed and cannot extend the embargo.

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan: Canada (2016-04-14): https://cdn.clinicaltrials.gov/large-docs/55/NCT01600755/Prot_SAP_000.pdf
  • Study Protocol and Statistical Analysis Plan: United Kingdom (2017-01-24): https://cdn.clinicaltrials.gov/large-docs/55/NCT01600755/Prot_SAP_001.pdf